CLINICAL TRIAL: NCT06679439
Title: A Prospective, Randomized Comparison of Dermis Vs. Auricular Cartilage Grafts for the Surgical Correction of Lower Eyelid Retraction
Brief Title: Comparison of Dermis Vs. Auricular Cartilage Grafts for the Surgical Correction of Lower Eyelid Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91414518.4.00000068
Record Dates: First submitted 2024-10-23; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Lower Eyelid Retraction
Keywords: eyelid; lower eyelid retraction

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cartilage graft group (Active Comparator): Patients with stable lower eyelid retraction that are submitted to surgical treatment using cartilage graft as spacer
  Interventions: Procedure: Surgical correction of lower eyelid retraction using autologous cartilage
- Dermis graft group (Active Comparator): Patients with stable lower eyelid retraction that are submitted to surgical treatment using dermis graft as spacer
  Interventions: Procedure: Surgical correction of lower eyelid retraction using autogenous dermis graft spacer.

INTERVENTIONS:
Procedure: Surgical correction of lower eyelid retraction using autologous cartilage — Surgical correction of lower eyelid retraction (LER) was performed using transcanthal cantopexy along with the insertion of an autogenous auricular cartilage graft spacer.
  Arms: Cartilage graft group
Procedure: Surgical correction of lower eyelid retraction using autogenous dermis graft spacer. — Surgical correction of lower eyelid retraction (LER) was performed using transcanthal cantopexy along with the insertion of an autogenous dermis graft spacer.
  Arms: Dermis graft group

SUMMARY:
This study aimed to compare the effectiveness of two autologous grafts-dermis and auricular cartilage-in the surgical correction of the lower eyelid retraction. Our primary focus was assessing changes in lower eyelid position using lower eyelid Margin to corneal Reflex Distance measurements, a.k.a Margin reflex distance 2 (MRD2).

DETAILED DESCRIPTION:
This prospective, randomized interventional study includes patients with stable LER. Patients are randomly assigned to undergo surgical correction using either auricular cartilage or dermis grafts, with the vertical dimension configured to be twice the scleral show height. MRD2 measurements were taken pre-operatively and at several post-operative intervals, with complications and outcomes recorded.

ELIGIBILITY:
Inclusion Criteria:

* eyelid retraction, scleral show

Exclusion Criteria:

* incomplete follow-up (less than 6 months), pregnancy and other abnormal ocular conditions or symptoms that preclude the patient's admission to the study, according to the clinical judgment of the investigator.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Lower eyelid Margin Reflex Distance measurements (MRD2) in millimeters | 6 months
  Data collected includes measurements of lower eyelid retraction using MRD2 from pre- and at 7 days, one month, three months, and six months' postoperative in facial frontal view photographs. Measurements are performed in a PC with Image J tool on digital photographs.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
our results will be published

REFERENCES:
- See also: Hospital site — https://www.hc.fm.usp.br/hc/ouvidoria/